CLINICAL TRIAL: NCT02508857
Title: Magnesium Sulfate Improves Postoperative Analgesia in Laparoscopic Gynecologic Surgeries: a Double-blind Randomized Controlled Trial.
Brief Title: Magnesium Sulfate Improves Postoperative Analgesia in Laparoscopic Gynecologic Surgeries
Acronym: Magnesium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NP0792010
Record Dates: First submitted 2015-04-27; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Pain, Postoperative
Keywords: pain, postoperative; anesthesia adjuvants; magnesium sulfate
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Magnesium; Magnesium Sulfate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ketorolac (Active Comparator): intravenous ketorolac (30 mg) is injected in bolus, followed by continuous infusion of saline solution (Group K) during the surgical procedure
  Interventions: Drug: Ketorolac
- magnesium (Experimental): intravenous magnesium sulfate (20 mg/kg) is injected in bolus, followed by continuous infusion of magnesium sulfate (2 mg/kg/h) (Group M) during the surgical procedure
  Interventions: Drug: Magnesium
- saline (Placebo Comparator): intravenous saline solution (20 ml) is injected in bolus, followed by continuous infusion of saline infusion during the entire procedure (Group S).
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Ketorolac — Patients received intravenous injection of ketorolac (30 mg) in bolus; then, saline solution was continuously infused during the entire procedure (Group K),
  Other Names: Toradol
  Arms: ketorolac
Drug: Magnesium — Patients received intravenous magnesium sulfate (20 mg/kg) in bolus, then magnesium sulfate (2 mg/kg/h) was continuously injected during the procedure (Group M)
  Other Names: Magnesium sulfate
  Arms: magnesium
Drug: Saline solution — intravenous saline solution (20 ml) was injected in bolus, followed by continuous infusion of saline solution during the entire procedure (Group S).
  Other Names: Sodium chloride
  Arms: saline

SUMMARY:
Magnesium sulfate has been reported to improve postoperative pain, but evidence is still controversial. Some studies demonstrated benefits while others concluded that there is no efficacy. Aim: the aim of the study was to compare the effect of intravenous infusion of magnesium sulfate to ketorolac during laparoscopic gynecologic oncology surgeries. Methods: We designed a double-blind randomized controlled trial that compared intravenous magnesium sulfate to ketorolac and saline solution in postoperative pain, morphine consumption and opioid related side effects.

DETAILED DESCRIPTION:
Sixty American Society of Anesthesiologists (ASA) I-II patients undergoing laparoscopic gynecologic oncology surgeries are enrolled in this study.

Patients were randomized to receive either intravenous ketorolac 30 mg in bolus followed by saline infusion (Group K), intravenous magnesium sulfate 20 mg/kg in bolus followed by magnesium 2 mg/kg/h (Group M) or intravenous saline solution 20 ml in bolus followed by saline infusion during the entire procedure (Group S). The study use a double-blinded methodology with random allocation into three groups using sealed opaque envelopes numbered 1 to 60, containing the instructions for the study. An independent anesthesiologist not involved in the study prepared the solutions and an observer who was also blinded to the patient's group records the data.

In the preoperative visit, patients that agree to participate are instructed about numeric rating scale (NRS) and the Patient Controlled Analgesia (PCA) device.

The night before surgery, patients are premedicated with midazolam 7.5 mg per os. Upon arrival in the operating room, monitoring devices (ECG, non-invasive arterial pressure, capnography, pulse oximetry) and a bispectral index (BIS) monitor are established. An intravenous line is secured, general intravenous anesthesia is induced with target infusion remifentanil and propofol. Cisatracurium besylate (0.5 mg/kg) is given to facilitate tracheal intubation and controlled ventilation is adjusted to maintain normocapnia with a 50% oxygen fraction administered. Then, the study medications are administered in bolus during 20 minutes, followed by continuous infusion of the specific solution, according to the study group to which the patient belonged, as described before.

At the end of the surgery, the study drugs are discontinued before the patient is extubated. If patients present clinical signs of residual neuromuscular blockade, they receive atropine 0.01mg/kg and neostigmine 0.04mg/kg. All patients receive dipyrone 30 mg/kg in bolus and a PCA device is connected to the intravenous line before discharge to the Post Anesthesia Care Unit (PACU). PCA solution containing morphine 1mg/ml in 0.9% saline, is set to give bolus of 2ml (2mg) with a 10min lockout interval.

In the postoperative period, the anesthesiologist responsible for the study question the intensity of pain in the patients using two methods: numerical rating scale (NRS) (0=no pain and 10=worst pain imaginable) and descriptive verbal scale (no pain, mild pain, moderate pain or severe pain - at emergence from anesthesia and after 20, 30 and 60 minutes, while in PACU. Patients are instructed to use the PCA device whenever they feel pain. Agitation and Sedation are monitored using RASS scale and patient is considered sedated if RASS ≤ -1. Episodes of nausea, vomiting, respiratory depression or pruritus are also recorded.

Patients are discharged to the ward after 60 minutes, if minimum criteria for discharge are met.

Time (in minutes) to the first morphine rescue, and total consumption of morphine in PACU are registered. After 24 hours, pain intensity score, total morphine consumption and side effects are also recorded and PCA device is disconnected.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II female patients undergoing laparoscopic gynecologic oncology surgeries, for treatment of cancer

Exclusion Criteria:

* chronic pain, cardiovascular, hepatic or renal disease, neuromuscular disease, diabetes, drugs or alcohol abuse, obesity, patients treated with calcium channel blockers or magnesium, allergy or contraindication to any of the drugs studied.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 24 hours
  intensity of pain in the patients using numerical rating scale (NRS) (0=no pain and 10=worst pain imaginable) and descriptive verbal scale (no pain, mild pain, moderate pain or severe pain

SECONDARY OUTCOMES:
time to first morphine rescue | first 6 hours
  Time (in minutes) to the first dose of morphine
morphine consumption | 60 minutes
  total consumption of morphine in PACU

CONTACTS AND LOCATIONS:
Overall Officials: angela m sousa, phD, Principal Investigator — Cancer Institute of the State of Sao Paulo
Locations (1):
- Angela Maria Sousa, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Result] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270